CLINICAL TRIAL: NCT05527912
Title: A Single-arm、Multicenter、Open-label、Phase II Clinical Study of the Combination of Rituximab、Chidamide、Zanubrutinib-induced and CHOP Therapy for Untreated Dual-expressing Diffuse Large B Cell Lymphoma
Brief Title: A Phase II Study of Rituximab, Chidamide, Zanubrutinib-induced and CHOP Therapy
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Li Zhiming, LiZhiming, Sun Yat-sen University
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: B2022-588-01
Record Dates: First submitted 2022-08-30; First posted 2022-09-06 (Actual); Last update posted 2023-04-25 (Actual); Status verified 2023-04

CONDITIONS: Double Express Diffuse Large B-cell Lymphoma
MeSH Terms: interventions — Rituximab; N-(2-amino-5-fluorobenzyl)-4-(N-(pyridine-3-acrylyl)aminomethyl)benzamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Arm I (RCZ WITH CHOP) (Experimental): Rituximab, Chidamide, Zanubrutinib-induced and CHOP Therapy
  Interventions: Drug: Rituximab, Chidamide, Zanubrutinib-induced and CHOP Therapy

INTERVENTIONS:
Drug: Rituximab, Chidamide, Zanubrutinib-induced and CHOP Therapy — All subjects received two courses of the following treatment:
  Rituximab ，375mg/m²， D1； Chidamiade ，20mg ，biw， d1-14； Zanubrutinib ，160mg， bid， d1-21；
  three weeks for a period of treatment, all subjects complete tumor assessment after two courses of treatment, patients which achieve complete remission continue for up to 8 sessions, patients achieve partial response and stable disease combined use of the following CHOP threapy to 6 courses, Patients with progressive disease dropped out of this research.
  CHOP Therapy:
  Cyclophosphamide， 750mg/m² ，D1； Vincristine， 1.4mg/m² ，D1 (maximum：2mg)； Doxorubicin or pirarubicin， 50mg/m²， D1； Prednisone ，30mg ，tid， D1-5.
  Other Names: RCZ WITH CHOP

SUMMARY:
This phase II trial studies how well giving rituximab,chidamide, and zanubrutinib with Sequential chemotherapy works in treating patients with double express diffuse large B-cell lymphoma. The prognosis of patients with DEL-DLBCL is usually worse than that of ordinary DLBCL.

ELIGIBILITY:
Inclusion Criteria:

1. Newly diagnosed dual-expression diffuse large B-cell lymphoma (DLBCL) with IHC BCL2 expression ≥50% and MYC expression ≥40%.
2. Male or female patients: 18-65 years old.
3. ECOG physical status score: 0~2 points.
4. Estimated survival time ≥6 months.
5. There must be at least 1 evaluable or measurable lesion that meets Lugano 2014 criteria [ evaluable lesion : 18F-fluorodeoxyglucose/Positron Emission Tomography (18FDG/PET) examination showed elevated lymph node or extranodal local uptake (higher than liver) and PET and/or Computed Tomography (CT) features consistent with lymphoma. Measurable lesion : Nodules >15mm or extranodal lesions >10mm with increased 18FDG uptake]. The absence of measurable lesions and increased diffuse hepatic uptake of 18FDG should be excluded.
6. Major organ function was good, that is, the following requirements should be met one week before enrollment: blood routine, WBC≥3×10*9/L, Hb≥80g/L,PLT≥80×10*9/L; The heart and liver functions were normal (TBIL≤1.5ULN, ALT and AST ≤2.5ULN), renal function was normal (1.5 times serum Cr≤1.5ULN), and no coagulation abnormalities were observed.
7. LVEF≥50% by echocardiography.
8. Women of childbearing age must have a pregnancy test (serum or urine) with a negative result within 14 days before enrollment and be willing to use a reliable method of contraception during the trial.
9. Subjects volunteered to join the study, signed informed consent, had good compliance, and cooperated with follow-up.

Exclusion Criteria:

1. Special types of DLBCL: DLBCL associated with chronic inflammation, lymphomatoid granuloma, primary mediastinal large B-cell lymphoma, B-cell lymphoma that cannot be classified (with intermediate features between DLBCL and classical Hodgkin's lymphoma), and primary central nervous system (CNS) DLBCL.
2. Transformed DLBCL (such as follicular lymphoma, chronic lymphocytic leukemia/small B-cell lymphoma transformed DLBCL), secondary central nervous system invasion of DLBCL.
3. A history of malignancies other than squamous cell carcinoma of the skin, basal cell carcinoma of the skin, or carcinoma in situ of the cervix within the past 5 years.
4. Major surgical procedures (excluding diagnostic procedures) performed within the past 2 months.
5. Previous NHL treatment: including chemotherapy, immunotherapy, radiotherapy, monoclonal antibody therapy, surgical treatment (except diagnostic surgery and biopsy).
6. Previous treatment with cytotoxic drugs or mab CD20 antibodies for other diseases (e.g., rheumatoid arthritis).
7. Those who used any monoclonal antibody within 3 months before enrollment, participated in other clinical trials and used other trial-related drugs, and were vaccinated with (attenuated) live virus vaccine within 1 month before enrollment.
8. Had used hematopoietic cytokines within 2 weeks before enrollment.
9. Patients with suspected active or latent tuberculosis.
10. Personswith known active bacterial, viral, fungal, mycobacterial, parasitic, or other infections (excluding fungal infections of the nail bed skin) or any major systemic infection event requiring intravenous antibiotic treatment or hospitalization within 4 weeks prior to enrollment (except neoplastic fever) .
11. Hiv-positive persons. Active HBV-positive and HCV-positive individuals, but those whose disease was judged to be under control, should be enrolled with caution, but should undergo effective antiviral intervention.
12. Other serious medical conditions that may limit the subject's participation in the study, such as uncontrolled diabetes; Severe cardiac insufficiency (NYHA grade II or above); Acute coronary syndrome in the last 6 months; Coronary revascularization such as stenting, cabG, and other cardiac and macrovascular procedures within the last 6 months; Severe arrhythmias include frequent ventricular premature, ventricular tachycardia, rapid atrial fibrillation/flutter, and severe bradycardia. （Uncontrolled hypertension: greater than 150/100mmHg). Gastric ulcers (those identified by the investigators as being at risk for perforation); Active autoimmune diseases; Severe hypertension; Patients with severe respiratory disease (e.g., obstructive pulmonary disease and history of bronchospasm), such as patients with a known history of interstitial pneumonia or a high suspicion of interstitial pneumonia; Or may interfere with the detection or management of suspected drug-related pulmonary toxicity.
13. Contraindications for any of the study drugs, including previous anthracyclines; Patients with diabetes who could not tolerate prednisone in this protocol.
14. Subject has a history of alcohol or drug abuse.
15. Persons with allergies or known allergies to any pharmaceutical active ingredient, excipient, or murine product or xenogeneic protein included in this test.
16. People with severe mental illness.
17. Patients who were unable to comply during the trial and/or follow-up phase.
18. Patients unable to swallow the study drug properly. Those who were deemed ineligible by the researchers.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2023-02-24 (Actual); Primary Completion 2024-09-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
EOT-CRR | 12 months
  End of Treatment Complete Response Rate

SECONDARY OUTCOMES:
EOT-ORR | 12 months
  End of Treatment Overall Response Rate
EOT-CRR2 | 2 months
  End of Initial two courses of Treatment Complete Response Rate
2year-PFS | 24 months
  2-year Progression Free Survival Rate
2year-OS | 24 months
  2-year Overall Survival Rate

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Department of Medical Oncology,Sun Yat-Sen University Cancer Center, Guangzhou, Guangdong
  - Sun Yat-sen University Cancer Center, Guangzhou

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP